CLINICAL TRIAL: NCT02185911
Title: Observational Study of Correction of Anaemia With Darbepoetin Alfa at Monthly Dose Frequency in EU and Australian Patients With Chronic Kidney Disease Not on Dialysis
Brief Title: Observational Study of Correction of Anaemia With Darbepoetin Alfa at QM Dosing Interval in Patients With CKD Not on Dialysis
Acronym: ADAPTATION
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20130301
Record Dates: First submitted 2014-06-26; First posted 2014-07-10 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Anaemia; Chronic Kidney Disease (CKD)
Keywords: chronic kidney disease,; anaemia correction/maintenance,; non dialysis,
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with CKD

SUMMARY:
To describe anaemia correction via haemoglobin measurements taken throughout observation period in ESA naive patients with chronic kidney disease initiated on darbepoetin alfa QM

DETAILED DESCRIPTION:
Darbepoetin alfa (Aranesp) is a long-acting ESA approved for treatment of anaemia in CKD patients, and may be administered once a week (QW), once every two weeks (Q2W) or once a month (QM) for correction and for maintenance in CKD patients not on dialysis. Prescribing information for darbepoetin alfa was updated in August 2013 (in EU and Australia), to incorporate the option for correction at QM dosing frequency in CKD patients not on dialysis. There is very little published literature describing QM correction in a real-world setting.

Data obtained from this study are intended to contribute to filling a literature gap and to provide a robust source of information for physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age.
2. Patients with CKD:

   1. Not on dialysis at time of darbepoetin alfa initiation at QM dosing frequency.
   2. Hb <10g/dL immediately prior to initiation of darbepoetin alfa at QM dosing.
   3. Commenced darbepoetin alfa at QM dosing frequency during or after August 2013.
   4. Received at least three consecutive doses of darbepoetin alfa at QM dosing frequency, being the initiation dose and two further doses at QM dosing frequency.
3. Patient or patient's legally acceptable representative has provided informed consent, if applicable according to local requirements.

Exclusion Criteria:

1. Treatment with an ESA within 14 weeks prior to initiation of darbepoetin alfa.
2. Patient was enrolled in an interventional device or drug study at any time during the 46-week data observation period or within 30 days prior to commencement of the data observtion period.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises CKD patients not on dialysis, ESA-naïve at time of initiation of darbepoetin alfa QM, and treated at nephrology clinics in EU and Australia from 01 May 2013. Eligible patients will have received at least three consecutive doses of darbepoetin alfa for correction of anaemia at a QM dosing interval. At each participating study site, all potentially elgible patients are to be considered for enrolment.
Sampling Method: Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Monthly Haemoglobin values | During the 32 weeks post initiation of darbepoetin alfa QM
  Monthly Hb within 10-12g/dL during the 32 weeks post initiation of darbepoetin alfa QM

SECONDARY OUTCOMES:
Doses of darbepoetin alfa/other ESAs over time | Throughout the 46 week observation period
  Doses of darbepoetin alfa/other ESAs over time (dose, route, frequency)
Haemoglobin values | Throughout the 46 week observation period
  Haemoglobin over the observation period
Change in Haemoglobin values | Throughout the 46 week observation period
  Change in haemoglobin from baseline
Increase in haemoglobin from baseline | Throughout the 46 week observation period
  Increase in haemoglobin of at least 1g/dL from baseline
Haemoglobin excursions | Throughout the 46 week observation period
  Haemoglobin excursions (<10,>12 g/dL) over the observation period
First haemoglobin within 10-12g/dL | During the 32 weeks post initiation of darbepoetin alfa QM
  Time from initiation of darbepoetin alfa QM to first haemoglobin within 10-12g/dL
first dose frequency change after third dose of darbepoetin alfa QM | During the 32 weeks post initiation of darbepoetin alfa QM
  Time from third dose of darbepoetin alfa at QM dosing frequency to first frequency change
Subjects remaining on darbepoetin alfa QM | During the 32 weeks post initiation of darbepoetin alfa QM
  Remaining on darbepoetin alfa QM for the full 32 weeks post initiation
TSAT, ferritin and albumin values | Throughout the 46 week observation period
  TSAT, ferritin and albumin over the observation period
Iron Use | Throughout the 46 week observation period
  Iron use (dose/route) over the observation period
Transfusions | Throughout the 46 week observation period
  Transfusions over the observation period (number of tranfusions and the number of units transfused)
Hospitalisations | Throughout the 46 week observation period
  Hospitalisations (duration and primary cause) over the observation period

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (33):
- Austria (3):
  - Research Site, Feldkirch
  - Research Site, Linz
  - Research Site, Vienna
- Bulgaria (7):
  - Research Site, Dobrich
  - Research Site, Montana
  - Research Site, Pazardzhik
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Vratsa
- Czechia (4):
  - Research Site, Brno
  - Research Site, Havlíčkův Brod
  - Research Site, Nové Město na Moravě
  - Research Site, Třebíč
- Greece (3):
  - Research Site, Athens
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Baja
  - Research Site, Kecskemét
  - Research Site, Szeged
  - Research Site, Szigetvár
  - Research Site, Szombathely
  - Research Site, Zalaegerszeg
- Research Site, Albano Laziale RM, Italy
- Poland (5):
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Sieradz
  - Research Site, Stalowa Wola
- Spain (4):
  - Research Site, Córdoba, Andalusia
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Valencia, Valencia

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com